CLINICAL TRIAL: NCT06604832
Title: Effects of PrabotulinumtoxinA-xvfs on Facial Skin Quality, Fine Wrinkles, and Texture
Brief Title: Effects of Microtox on Facial Skin Quality, Fine Wrinkles, and Texture
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kalpna Kay Durairaj, MD, FACS (Other)
Collaborators: Evolus, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Kalpna Kay Durairaj, MD, FACS, Principal Investigator, K. Kay Durairaj, MD, FACS, A Medical Corporation
Organization: K. Kay Durairaj, MD, FACS, A Medical Corporation (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KDEJ24
Record Dates: First submitted 2024-09-17; First posted 2024-09-20 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Skin Aging; Skin Wrinkling
Keywords: Microtox; Minimally invasive; Skin quality; Skin texture; Fine wrinkling; Botulinum toxin; PrabotulinumtoxinA-xvfs; Glabellar lines
MeSH Terms: interventions — prabotulinumtoxin A; incobotulinumtoxinA; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treated with prabotulinumtoxinA-xvfs and placebo (Placebo Comparator): Subjects will have one treatment session at week 0 and two live assessment visits at weeks 2 and 12. Approximately 20 units of prabotulinumtoxinA-xvfs will be injected into the left side of the subject's glabellar lines and forehead region, and a placebo saline treatment will be injected into the right side of the subject's glabellar lines and forehead region.
  Interventions: Drug: PrabotulinumtoxinA-Xvfs; Drug: saline solution (placebo)
- Treated with prabotulinumtoxinA-xvfs and incobotulinumtoxinA (Active Comparator): Subjects will have one treatment session at week 0 and two live assessment visits at weeks 2 and 12. Approximately 20 units of prabotulinumtoxinA-xvfs will be injected into the left side of the subject's glabellar lines and forehead region, and approximately 20 units of incobotulinumtoxinA will be injected into the right side of the subject's glabellar lines and forehead region.
  Interventions: Drug: PrabotulinumtoxinA-Xvfs; Drug: IncobotulinumtoxinA

INTERVENTIONS:
Drug: PrabotulinumtoxinA-Xvfs — Each vial of prabotulinumtoxinA-xvfs contains 100 units of product, and it will be reconstituted with 5 mL of bacteriostatic saline solution. 20 units of this intervention will only be injected to the left side of subject faces - intramuscularly to the corrugator supercilii and intradermally to the forehead region.
  Other Names: Jeuveau
Drug: IncobotulinumtoxinA — Each vial of incobotulinumtoxinA contains 100 units of product, and it will be reconstituted with 5 mL of bacteriostatic saline solution. 20 units of this intervention will only be injected to the right side of subject faces - intramuscularly to the corrugator supercilii and intradermally to the forehead region.
  Other Names: Xeomin
  Arms: Treated with prabotulinumtoxinA-xvfs and incobotulinumtoxinA
Drug: saline solution (placebo) — As a placebo treatment, saline solution will be injected on the right side of the glabellar lines and forehead region instead of an active neuromodulator. The saline solution has no therapeutic effect and is used as a control to compare the results against the active treatment.
  Arms: Treated with prabotulinumtoxinA-xvfs and placebo

SUMMARY:
The goal of this split-face clinical trial is to test the efficacy of microtox in improving facial skin quality, fine wrinkles, and texture. Participants will:

* be randomly assigned to Group A (which will receive 20 units of neuromodulator on the left side of the forehead and a placebo saline treatment on the right side) or Group B (which will receive 20 units of neuromodulator on the left side of the forehead and 20 units of a different neuromodulator brand on the right side as a comparator)
* have one treatment session at week 0, and two live assessment visits at weeks 2 and 12
* have their pictures taken at each visit to track progress

DETAILED DESCRIPTION:
Twenty (20) subjects will be enrolled in the study. The subjects will have one treatment session at week 0, and two live assessment visits at weeks 2 and 12. Office visits will last approximately 2 hours. All subjects will have their photographs taken at the beginning of each visit to track progress. Photographs will be taken of the forehead in a relaxed state, with eyebrows furrowed, and with eyebrows raised. All pictures will be taken via the Quantificare LifeViz Micro and will be stored via a HIPAA-compliant server.

Subjects will be randomly assigned to one of two groups. Group A will receive 10 units of prabotulinumtoxinA-xvfs delivered intramuscularly to the corrugator supercilii on the left of the glabellar lines, 10 units of prabotulinumtoxinA-xvfs delivered intradermally (~1 mm depth) to the left side of the forehead region, and a placebo saline treatment on the right side of the glabellar lines and forehead region. Group B will receive 10 units of prabotulinumtoxinA-xvfs delivered intramuscularly to the corrugator supercilii on the left of the glabellar lines, 10 units of prabotulinumtoxinA-xvfs delivered intradermally (~1 mm depth) to the left side of the forehead region, and 20 units of incobotulinumtoxinA on the right side (intramuscularly in the glabellar region and intradermally in the forehead region.

100 units of botulinum toxin A will be reconstituted with 5 mL of bacteriostatic saline. After subjects have their picture taken, topical Lidocaine/Tetracaine 23%/7% ointment cream will be applied to the treatment sites. After 15 minutes of numbing, the topical anesthetic will be cleaned off with alcohol. Subjects will be asked to repeatedly furrow and raise their eyebrows to let the treating physician assess the muscle of interest. With the subject in a semi-reclined position, the treating physician will inject microboluses using a standard 30 gauge 0.5" needle.

At each visit, the treating physician will rate each subject according to the Scientific Assessment Scale of Skin Quality (SASSQ). The Global Aesthetic Improvement Scale (GAIS) will be used by the treating physician and subjects to rate aesthetic improvement at each visit after baseline. Subjects will also rate their overall aesthetic improvement and treatment satisfaction at each visit after baseline according to a 5-point scale: (1) Extremely dissatisfied, (2) Dissatisfied, (3) Slightly satisfied, (4) Satisfied, (5) Extremely satisfied. Before and after photos of treated patients will be independently evaluated by the blinded, secondary evaluator using the SASSQ scale at each time interval of photos taken.

ELIGIBILITY:
Inclusion Criteria:

* Biological females, 18-65 years old, of any race and ethnic background
* Individuals with mild to moderate facial wrinkles
* All skin types (Fitzpatrick I-VI)
* Willingness to participate and provide written informed consent
* Ability to follow study instructions and likely to complete all required visits

Exclusion Criteria:

* Females who are pregnant, breastfeeding, chronically using nonsteroidal anti-inflammatory drugs, have autoimmune conditions or have a known allergy to the study medications.
* Previous cosmetic procedures near the forehead within the last 6 months or botulinum toxin treatments within the last 4 months
* Known neuromuscular disorders or a hypersensitivity to botulinum toxin
* Significant dermatological conditions affecting the face
* Use of medications affecting neuromuscular function or skin healing within 2 weeks prior to the beginning of study
* Subject has a condition or is in a situation which, in the opinion of the Investigator, may put the subject at significant risk, may confound the study results, or may interfere significantly with participation in the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility is determined by their biological sex, as there are distinct physiological differences between male and female skin. Due to these differences, individuals whose gender identity differs from their biological sex (i.e., transgender individuals) are excluded from the study to ensure consistency in data collection related to sex-specific skin characteristics.
Enrollment: 20 (Actual)
Dates: Start 2024-09-03 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
Scientific Assessment Scale of Skin Quality (SASSQ) Rating | Up to 12 weeks
  The treating physician and the blinded, secondary evaluator will rate the subject after the final treatment. The scale identifies 6 parameters of skin quality: (1) loss of elasticity, (2) wrinkles, (3) roughness, (4) pigmentation/lentigines, (5) erythema, and (6) pore size. The scale has 5 points to describe the intensity of parameters 1-5: 0 implies none, 1 implies mild, 2 implies moderate, 3 implies severe, and 4 implies very severe. For parameter 6, 0 implies fine, 1 implies small, 2 implies moderate, 3 implies large, and 4 implies very large.
Global Aesthetic Improvement Scale (GAIS) Rating | Up to 12 weeks
  The treating physician and the blinded, secondary evaluator will rate the subject after the final treatment. Based on aesthetic appearance, qualitative success of treatment will be evaluated using the GAIS. Aesthetic appearance will be rated one of the five following options: - Worse: The appearance is worse than the original condition - No Change: The appearance is essentially the same as the original condition - Improved: Obvious improvement in appearance from the initial condition, but a touchup or re-treatment is indicated - Much Improved: Marked improvement in appearance but not completely optimal for this patient. A touchup would slightly improve the result - Very Much Improved: Optimal cosmetic result for the treatment in this patient.

SECONDARY OUTCOMES:
Scientific Assessment Scale of Skin Quality (SASSQ) Rating | Up to 2 weeks
  The treating physician and the blinded, secondary evaluator will rate the subject at each treatment visit using the SASSQ rating. The scale identifies 6 parameters of skin quality: (1) loss of elasticity, (2) wrinkles, (3) roughness, (4) pigmentation/lentigines, (5) erythema, and (6) pore size. The scale has 5 points to describe the intensity of parameters 1-5: 0 implies none, 1 implies mild, 2 implies moderate, 3 implies severe, and 4 implies very severe. For parameter 6, 0 implies fine, 1 implies small, 2 implies moderate, 3 implies large, and 4 implies very large.
Global Aesthetic Improvement Scale (GAIS) Rating | Up to 2 weeks
  Based on aesthetic appearance, qualitative success of treatment will be evaluated by the treating physician and the blinded, secondary evaluator using the GAIS. Aesthetic appearance will be rated one of the five following options: - Worse: The appearance is worse than the original condition - No Change: The appearance is essentially the same as the original condition - Improved: Obvious improvement in appearance from the initial condition, but a touchup or re-treatment is indicated - Much Improved: Marked improvement in appearance but not completely optimal for this patient. A touchup would slightly improve the result - Very Much Improved: Optimal cosmetic result for the treatment in this patient
Global Aesthetic Improvement Scale (GAIS) Rating | Up to 12 weeks
  Based on aesthetic appearance, qualitative success of treatment will be self-evaluated by subjects using the GAIS. Aesthetic appearance will be rated one of the five following options: - Worse: The appearance is worse than the original condition - No Change: The appearance is essentially the same as the original condition - Improved: Obvious improvement in appearance from the initial condition, but a touchup or re-treatment is indicated - Much Improved: Marked improvement in appearance but not completely optimal for this patient. A touchup would slightly improve the result - Very Much Improved: Optimal cosmetic result for the treatment in this patient
Scientific Assessment Scale of Skin Quality (SASSQ) Rating | Up to 12 weeks
  Based on aesthetic appearance, qualitative success of treatment will be self-evaluated by subjects using the SASSQ. The scale identifies 6 parameters of skin quality: (1) loss of elasticity, (2) wrinkles, (3) roughness, (4) pigmentation/lentigines, (5) erythema, and (6) pore size. The scale has 5 points to describe the intensity of parameters 1-5: 0 implies none, 1 implies mild, 2 implies moderate, 3 implies severe, and 4 implies very severe. For parameter 6, 0 implies fine, 1 implies small, 2 implies moderate, 3 implies large, and 4 implies very large.
Patient Satisfaction with Treatment and Aesthetic Appearance | Up to 12 weeks
  Subjects will rate their satisfaction at each visit. Patient satisfaction will be assessed using a 5-point scale: (1) extremely dissatisfied, (2) dissatisfied, (3) slightly satisfied, (4) satisfied, and (5) extremely satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Kalpna K Durairaj, MD, Principal Investigator — K. Kay Durairaj, MD, A Medical Corp.
Locations (1):
- K. Kay Durairaj, MD, A Medical Corp., Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with interest in microtox and its effect on facial skin quality. Individual participant data that underlies the results reported in this article will be shared after identification. Approval of the request and execution of all applicable agreements (e.g., a material transfer agreement) are prerequisites to the sharing of data with the requesting party. Furthermore, the proposed use of trial IPD must be approved with an Independent Review Committee prior to any data sharing.
Supporting Information: Study Protocol
Time Frame: Data will become available beginning 12 months and ending 28 months after article publication. Upon approval of a data sharing request, data will be accessible to researchers for up to 3 months.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in scientific research, and will be provided following review and approval of a research proposal, Statistical Analysis Plan (SAP), and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact research@beautybydrkay.com.

REFERENCES:
- [Background] Hanna E, Xing L, Taylor JH, Bertucci V. Role of botulinum toxin A in improving facial erythema and skin quality. Arch Dermatol Res. 2022 Oct;314(8):729-738. doi: 10.1007/s00403-021-02277-0. Epub 2021 Sep 14. PMID 34519860
- [Background] Shin DM, Lee J, Noh H, Jang D, Oh SJ, Park JH, Lee JH. A Double-Blind, Split-Face, Randomized Study on the Effects and Safety of Intradermal Injection of Botulinum Toxin A (Incobotulinum Toxin A) in the Cheek. Ann Dermatol. 2022 Dec;34(6):442-450. doi: 10.5021/ad.21.316. PMID 36478426
- [Background] Shuo L, Ting Y, KeLun W, Rui Z, Rui Z, Hang W. Efficacy and possible mechanisms of botulinum toxin treatment of oily skin. J Cosmet Dermatol. 2019 Apr;18(2):451-457. doi: 10.1111/jocd.12866. Epub 2019 Jan 29. PMID 30697928
- [Background] Eiben-Nielson C, Kerscher M. Development and validation of a global photonumeric scale for evaluating skin quality of aged female facial skin. J Cosmet Dermatol. 2021 Dec;20(12):4032-4039. doi: 10.1111/jocd.14058. Epub 2021 Mar 24. PMID 33690945
- [Background] Park JY, Cho SI, Hur K, Lee DH. Intradermal Microdroplet Injection of Diluted Incobotulinumtoxin-A for Sebum Control, Face Lifting, and Pore Size Improvement. J Drugs Dermatol. 2021 Jan 1;20(1):49-54. doi: 10.36849/JDD.5616. PMID 33400411
- [Background] Fabi SG, Park JY, Goldie K, Wu W. Microtoxin for Improving Pore Size, Skin Laxity, Sebum Control, and Scars: A Roundtable on Integrating Intradermal Botulinum Toxin Type A Microdoses Into Clinical Practice. Aesthet Surg J. 2023 Aug 17;43(9):1015-1024. doi: 10.1093/asj/sjad044. PMID 36857534
- [Background] Diaspro A, Calvisi L, Manzoni V, Sito G. Microbotulinum: A Quantitative Evaluation of Aesthetic Skin Improvement in 62 Patients. Plast Reconstr Surg. 2020 Nov;146(5):987-994. doi: 10.1097/PRS.0000000000007248. PMID 33136941